CLINICAL TRIAL: NCT05655416
Title: Endovenous Chemical Ablation and Trendlenburg Operation for the Treatment of Great Saphenous Vein Varicosities
Brief Title: Treatment of Great Saphenous Vein Varicosities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Walied Khereba, Principal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endovenous chemical ablation
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lower limb varicose vein (Other)
  Interventions: Procedure: Endovenous chemical ablation with Trendelenburg's operation (eCAT)

INTERVENTIONS:
Procedure: Endovenous chemical ablation with Trendelenburg's operation (eCAT) — Endovenous chemical ablation with trendelenburg's operation (e CAT) is a method for the treatment of varicose veins

SUMMARY:
Venous insufficiency at lower extremities may result in clinical problems from cosmetic issues to ulcerations. When the frequency of venous insufficiency and its related problems are considered besides their diversity, it is encountered as a public health issue. This pathology is reported to affect 40% of women and 20% of men.1 Patients with varicose veins may complain of unsightly appearance, aching, heaviness, pruritus, and early fatigue of the affected leg. These symptoms worsen with prolonged standing and sitting and are relieved by elevation of the leg above the level of the heart. Also, mild edema is often present. More severe signs include thrombophlebitis, hyperpigmentation, lipodermatosclerosis, ulceration, and bleeding

ELIGIBILITY:
Inclusion Criteria:

* Patients presented by primary VV of the LL complaining of Leg pain cosmetic disfigurement, leg ulcer, itching, or pigmentation at LL
* the incompetence of the saphenofemoral junction (SFJ) and or saphenopopliteal junction (SPJ).

Exclusion Criteria:

* Lower limb involvement by any of the following conditions; secondary VV, recurrent VV, lymphedema, acute superficial thrombophlebitis, arterio-venous fistula (congenital or acquired), congenital anomalies of the venous system, general comorbidities, skin infection or ischemia

Ages: 20 Years to 60 Years | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
GSV Patency | at one week post operative
  Great saphenous Vein Patency: is a categorical outcome that will be assesd by dopler ultrasound. it may be patent or partilly occluded or completely occluded or recanalized.
GSV Patency | at one month post operative
  Great saphenous Vein Patency: is a categorical outcome that will be assesd by dopler ultrasound. it may be patent or partilly occluded or completely occluded or recanalized.
GSV Patency | at one year post operative
  Great saphenous Vein Patency: is a categorical outcome that will be assesd by dopler ultrasound. it may be patent or partilly occluded or completely occluded or recanalized.

CONTACTS AND LOCATIONS:
Locations (1):
- Walied Khereba, Zagazig, Egypt